CLINICAL TRIAL: NCT01397240
Title: The Safety and Efficacy of Albis®: The Prevention of Aspirin-induced Gastrointestinal Ulcers in Patients Taking Low-dose Aspirin, A Pilot Study
Brief Title: The Safety and Efficacy of Albis®: The Prevention of Aspirin-induced Gastrointestinal Ulcers in Patients
Acronym: AL-PA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DW_ABS002P
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2011-07

CONDITIONS: Patients Taking Low-dose Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albis (Experimental): Drug: Albis Tab 2 tab, twice a day
  Interventions: Drug: Albis Tab
- Placebo (Placebo Comparator): Placebo 2 tab, twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albis Tab — 2 Tab, twice a day, 12 weeks
  Arms: Albis
Drug: Placebo — 2 Tab, twice a day, 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to research the safety and efficacy of Albis® for the prevention of aspirin-induced gastrointestinal ulcers in patients taking low-dose aspirin.

DETAILED DESCRIPTION:
The Safety and Efficacy of Albis®: The Prevention of Aspirin-induced Gastrointestinal Ulcers in Patients taking Low-dose Aspirin, A pilot study Double-Blind, Placebo-Controlled, Randomized, Multicenter, Parallel, Prospective study

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 20 to 80 years
* Subjects identified with at least one of the following diagnosis (Angina, Myocardial Infarction(Old), Cerebrovascular Disease, Peripheral Vascular Disease, Diabetes, Hypertension, Hypercholeseterolemia, Obesity) who are required to take a low dose of Aspirin (100mg/day) for more than 12 weeks.

Exclusion Criteria:

* Females who are pregnant, nursing, or planning a pregnancy during the study period or females of childbearing potential
* Peptic ulcer or Reflux oesophagitis
* hemostatic disorder or coagulation disorder
* Known allergy or hypersensitivity to the study medication

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-01 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Gastric Ulcer | 2 years

SECONDARY OUTCOMES:
Incidence rate of gastiritis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Jin Park, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam severance Hospital, Seoul, South Korea